CLINICAL TRIAL: NCT04570865
Title: Dapagliflozin And Pulmonary Artery Hemodynamics in Heart Failure With Reduced Ejection Fraction Patients With CardioMEMS®
Acronym: DAPA-MEMS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Scripps Health (Other)
Responsible Party: Principal Investigator, James Thomas Heywood, Director of the Advanced Heart Failure Program, Scripps Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAPA-MEMS
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: The focus of this study is to investigate the use of Dapagliflozin in HFrEF (NYHA II-IV) patients with or without diabetes who have CardioMEMS® implanted to assess the impact on pulmonary artery pressure measurements after 12 weeks of therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Dapagliglozin (Experimental): The focus of this study is to investigate the use of Dapagliflozin in HFrEF (NYHA II-IV) patients with or without diabetes who have CardioMEMS® implanted to assess the impact on pulmonary artery pressure measurements after 12 weeks of therapy.
  Interventions: Drug: Dapagliflozin; Device: CardioMEMS

INTERVENTIONS:
Drug: Dapagliflozin — The focus of this study is to investigate the use of Dapagliflozin in HFrEF (NYHA II-IV) patients with or without diabetes who have CardioMEMS® implanted to assess the impact on pulmonary artery pressure measurements after 12 weeks of therapy.
Device: CardioMEMS — The focus of this study is to investigate the use of Dapagliflozin in HFrEF (NYHA II-IV) patients with or without diabetes who have CardioMEMS® implanted to assess the impact on pulmonary artery pressure measurements after 12 weeks of therapy.

SUMMARY:
The focus of this study is to investigate the use of Dapagliflozin in HFrEF (NYHA II-IV) patients with or without diabetes who have CardioMEMS® implanted to assess the impact on pulmonary artery pressure measurements after 12 weeks of therapy.

DETAILED DESCRIPTION:
Prior studies have demonstrated an association between the use of sodium-glucose cotransporter 2 (SGLT-2) inhibitors for diabetic patients and reductions in composite primary outcomes of cardiovascular mortality, nonfatal myocardial infarction, or nonfatal stroke, as well as reductions in heart failure among patients with diabetes. The 2019 DAPA-HF trial studied whether the addition of the SCLT-2 inhibitor dapagliglozin could benefit patients with heart failure with reduced ejection fraction (HFrEF), either with or without diabetes. Results indicated that that SGLT-2 inhibitors resulted in 4.9% absolute reduction in the cardiovascular death or worsening heart failure and a 2.3% absolute reduction in all-cause mortality in patients with and without diabetes. Dapagliflozin is FDA approved to reduce the risk of cardiovascular death or hospitalization in patients with HFrEF with or without Type 2 diabtes. The mechanisms of cardiovascular benefit remain unclear, however it is likely to be driven by a reduction in heart failure death given that rates of myocardial infarction were similar between treatment arms.

The CardioMEMS® system is an implantable device that can measure pulmonary artery systolic, diastolic and mean pressure on a daily basis. It has been shown convincingly that monitoring the MEMS device results in reduced pulmonary pressures and in turn a reduction in heart failure hospitalizations.

The focus of this study is to investigate the use of Dapagliflozin in HFrEF (NYHA II-IV) patients with or without diabetes who have CardioMEMS® implanted to assess the impact on pulmonary artery pressure measurements after 12 weeks of therapy.

ELIGIBILITY:
Inclusion Criteria

1. Diagnosis of HFrEF and existing CardioMEMs in place
2. Patients who have historically been compliant with CardioMEMS followup
3. Ejection fraction < or = to 40%
4. New York Heart Association (NYHA) class II-IV heart failure
5. Able to read and write in English Exclusion Criteria

1. creatinine clearance less than or equal to 45 2. History of renal transplant 3. systolic blood pressure less than 85 on time of initiation of drug 4. intolerance/allergy to farxiga 5. pregnant patients or those who are planning to become pregnant during the study period 6. unable to read and write in English 7. acutely hospitalized patients or those who were hospitalized in the past 30 days 8. history of noncompliance with CardioMEMS followup 9. History of frequent mycotic urinary tract infections 10. History of organ transplantation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Effect of Dapagliflozin on pulmonary diastolic pressure from baseline to 12 weeks of therapy Secondary End Points | 12 weeka
  PA diastolic pressure change
Compare the change in PA pressures, systolic and mean, from baseline to 12 weeks. | 12 weeks
  PA pressure changes

SECONDARY OUTCOMES:
Describe the change in NT-ProBNP from baseline to 12 weeks | 12 weeks
  NTproBNP change

OTHER OUTCOMES:
Compare total diuretic dose from baseline to 12 weeks. | 12 weeks
  diuretic dose
Determine the change in 6 min walk distance from baseline to 12 weeks | 12 weeks
  6 MWT
Compare the change in KCCQ from baseline to 12 weeks. | 12 weeks
  KCCQ
Change in renal function estimated GFR from baseline to 12 weeks | 12 weeks
  renal function
Change in weight baseline to 12 weeks | 12 weeks
  weight

CONTACTS AND LOCATIONS:
Locations (1):
- Scripps Clinic, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] 1. Neal B, Perkovic V, Mahaffey KW, et al. Canagliflozin and Cardiovascular and Renal Events in Type 2 Diabetes. N Engl J Med. 2017;377(7):644-657. doi:10.1056/NEJMoa1611925 2. Zinman B, Wanner C, Lachin JM, et al. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015;373(22):2117-2128. doi:10.1056/NEJMoa1504720 3. Wiviott SD, Raz I, Bonaca MP, et al. Dapagliflozin and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2019;380(4):347-357. doi:10.1056/NEJMoa1812389 4. McMurray JJV, Solomon SD, Inzucchi SE, et al. Dapagliflozin in Patients with Heart Failure and Reduced Ejection Fraction. N Engl J Med. 2019;381(21):1995-2008. doi:10.1056/NEJMoa1911303 5. Abraham WT, Adamson PB, Bourge RC, et al. Wireless pulmonary artery haemodynamic monitoring in chronic heart failure: A randomised controlled trial. Lancet. 2011;377(9766):658-666. doi:10.1016/S0140-6736(11)60101-3